CLINICAL TRIAL: NCT01179724
Title: Comparison of Proton Pump Inhibitor and H2 Receptor Blocker on Prevention of Bleeding From Iatrogenic Ulcer After Endoscopic Submucosal Dissection for Gastric Neoplasms: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center IRB, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-06-030
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2009-06

CONDITIONS: Delayed Bleeding
MeSH Terms: interventions — Proton Pump Inhibitors; Pantoprazole

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- high dose proton pump inhibitor (Experimental)
  Interventions: Drug: high dose proton pump inhibitor
- H2 receptor antagonist (Active Comparator)
  Interventions: Drug: H2RB

INTERVENTIONS:
Drug: high dose proton pump inhibitor — IV loading PPI before 2hr to conduct ESD, and IV 8mg/h continuous infusion within 48hr, and then 40mg oral pantoprazole for one month
  Other Names: pantoprazole
  Arms: high dose proton pump inhibitor
Drug: H2RB — IV 50mg loading H2 receptor antagonist before 2hr to conduct ESD, and IV 13mg/h continuous infusion within 48hr, and then 300mg oral H2 receptor antagonist for one month
  Other Names: curan
  Arms: H2 receptor antagonist

SUMMARY:
after endoscopic submucosal dissection(ESD) of early gastric cancer, conventional proton pump(PPI) inhibitors and H2 receptor antagonists have a controversial effect on preventing bleeding from artificial ulcers. the aim of this study was to investigate whether a stronger acid suppression (high dose PPI) more effectively prevents bleeding after ESD

ELIGIBILITY:
Inclusion Criteria:

* the patients who agreed informed consent
* gastric adenoma or early gastric cancer which is eligible for conventional ESD indication

Exclusion Criteria:

* recent drug history of PPI, H2 rector antagonist, bismuth and antibiotics within 4 weeks
* recent drug history of anticoagulant or antiplatelet agent within 7 days
* s/p subtotal gastrectomy
* recurred gastric adenoma or cancer
* pregnant or breast feeding patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
bleeding incidence after ESD | time to occur delayed bleeding within one month after ESD

SECONDARY OUTCOMES:
the size of healing ulcer after ESD | follow up endoscopy for the healing of iatrogenic ulcer after one month ESD

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea